CLINICAL TRIAL: NCT03995303
Title: HOMEFOOD Study - Home Delivered Food and Nutrition Therapy for Discharged Geriatric Hospital Patients
Acronym: HOMEFOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Responsible Party: Principal Investigator, Alfons Ramel, Professor, University of Iceland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UI-2018-HOMEFOOD
Record Dates: First submitted 2019-01-09; First posted 2019-06-24 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Malnutrition
Keywords: Malnutrition; Old adults; Home-delivered meals; NCP - Nutrition Care Process; Food
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCP and home-delivered meals (Active Comparator): Preventing malnutrition with NCP by a registered dietician and home-delivered meals
  Interventions: Other: NCP and home-delivered meals
- Current practice (No Intervention): Current practice after discharge from the University Hospital of Iceland.

INTERVENTIONS:
Other: NCP and home-delivered meals — The dietitian (Ph.D. student) will perform an individual nutritional assessment focusing on dietary intake, activity level and weight of each participant, as a basis for developing an individualized nutrition care plan consistent with estimated nutritional requirements and nutritional rehabilitation goals. Total fluid, energy- and protein requirements will be estimated for each patient. Giving the group free food to fulfill protein-and energy needs.
  Other Names: NCP and delivered meals
  Arms: NCP and home-delivered meals

SUMMARY:
Because of short hospital stays, and nutritional status worsening for geriatric patients, time to improve this is limited. It seems necessary to integrate nutritional support after discharge, to prevent the consequences of malnutrition on health and physical capability. This study tests whether nutrition support using NCP (Nutrition Care Process) (1) in combination with delivered meals designed for old adults, improves nutritional status, muscle strength, physical function, quality of life and rehospitalization and mortality rates after discharge, compared to currently used care (2 = control) along with historical data. Participants (N = 200), will be randomized into two groups, the intervention will last 24 weeks. A dietitian (Ph.D. student) visits participants in the intervention group 5 times during the study period. Outcome parameters will be measured before discharge from the hospital, at 12 weeks and at 24 weeks. Data on hospital readmission and mortality will be followed up at 6 months after the intervention.

Condition or disease: Malnutrition Intervention/treatment: NCP by a dietitian and free food constructed to fulfill protein and energy needs for the group.

DETAILED DESCRIPTION:
Malnutrition is common in older people admitted to the hospital and can worsen after discharge. Therefore, it seems necessary to integrate nutritional support not only during the hospital stay but also in the period after discharge. The aim of this Randomized Controlled Trial (RCT) is to test whether nutritional support provided by a dietitian, using Nutrition Care Process in combination with delivered meals designed for the needs of older adults (group 1), improves nutritional status, muscle strength, physical function, quality of life and as a secondary outcome re-hospitalization and/or mortality of geriatric patients with malnutrition risk after discharge compared to currently used standard care (group 2 = control).

Time and work plan:

After 12 months

* Need identification and product ideas ready
* Packaging material ready
* Estimate of the feasibility of meals for old adults
* Allowances from the ethical committee, the data protection committee, the Ph.D. committee of the Faculty of Food Science and Nutrition at the University of Iceland.

After 24 months

* The last participant recruited
* End of intervention

After 36 months

* End of follow up
* Database ready
* First paper submitted

Methods-Intervention

This 24-week randomized controlled trial will randomize the participants (N = 200) to two groups. The dietitian (Ph.D. student) will perform a total of 5 home visits during the study period to participants in the intervention group. Meals will be delivered weekly to the participants. Outcome parameters will be measured just before discharge from the hospital and after 12 weeks and at 24 weeks in the home of the participants. Data on hospital re-admission and mortality will also be followed up at 12 months.

The aim of the intervention is to implement individual dietetic advice and optimize participants' nutritional status by following the Nutritional Care Process*, involving nutritional assessment, diagnosis, intervention, monitoring, and evaluation. Dietary counseling, motivation, and education will help to maintain participants' body weight, and ensure that energy and protein requirements as well as for other critical nutrients are achieved.

*The Nutrition Care Process (NCP) reflects the current state of the art in nutrition care and is designed to improve the consistency and quality of individualized care for patients and the predictability of the patient outcomes. It is not intended to standardize nutrition care for each patient, but to establish a standardized process for providing care.

To achieve the aim, the dietitian (Ph.D. student) will meet the participants in the intervention group, six times.

* The day before discharge where baseline measurements will be done,
* 1 week after discharge,
* 3 weeks after discharge,
* 6 weeks after discharge,
* 9 weeks after discharge, and
* 12 weeks after discharge where endpoint measurements will be done. The dietitian (Ph.D. student) will perform an individual nutritional assessment focusing on dietary intake, activity level and weight of each participant, as a basis for developing an individualized nutrition care plan consistent with estimated nutritional requirements and nutritional rehabilitation goals. Total fluid, energy- and protein requirements will be estimated for each patient. To assess dietary intake, the dietitian will perform a dietary history interview at each visit to determine fluid, energy and protein intake of the participant. Strategies for achieving fluid, energy and protein requirements and achieving compliance included dietary counseling with attention to nutritional risk factors, timing, size and frequency of meals, recommendations for nutrient dense foods and drinks, and provision of educational material.

If relevant, the dietitian will:

* initiate the prescription of oral nutritional supplements with high energy and protein density that will be reimbursed by Health Insurance.
* Contact providers of meals-on-wheels to change the meals to high energy and protein dense menu or to mashed/puréed food.
* Recommend use of vitamin D, calcium and other vitamins-minerals considered necessary to achieve optimal nutritional status,
* Invite home care and community nursing staff to participate in home visits to achieve the best possible outcome for the patient by interdisciplinary collaboration.

If considered relevant the participants will receive a short consultation by telephone by the dietitian to give advice and to stimulate compliance to the proposed nutritional care plan in-between the home visits.

The control group will meet the dietitian/staff for baseline, 12 weeks and at the 24-week endpoint measurements. The control group will not receive any dietary counseling or education during the study period which reflects current clinical practice.

The Ph.D. students' contributions A Ph.D. student in clinical nutrition (Berglind Soffía Blondal) will be the project manager of the intervention study on a day-to-day base. The student will be supervised by Prof. Alfons Ramel and Assoc. Prof. Ólöf Guðný Geirsdóttir, both on the Faculty of Food Science and Nutrition. The student will be involved in application work to the ethical committee, screening, conduct of the intervention study, data work and writing of scientific papers.

Ethics The study has been approved by the Ethics Committee of Landspitali- University Hospital of Iceland and informed written consent will be obtained from all participants. The study can only improve the nutritional status of geriatric patients that take part in the intervention groups. The participants in the control group, however, won't get any nutritional interventions and therefore have a greater risk of re-admissions and a worse overall outcome compared to the intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the geriatric units at the University Hospital of Iceland discharging home to independent living
* A score of 20 or above on the Mini-Mental State Evaluation (MMSE) form
* Being at nutritional risk according to the validated nutritional risk screening tool (NRS-2002, score 3+)
* The capability of eating orally

Exclusion Criteria:

* Living at a nursing home
* MMSE score of under 20
* No nutritional risk

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Body weight | Measurement at discharge, baseline
  Body weight in kilograms
Body weight | Measurement at 12 weeks
  Body weight in kilograms
Body weight | Measurement at 24 weeks
  Body weight in kilograms
Five Times Sit to Stand Test | Measurement at discharge, baseline
  Part of short physical performance battery, yes vs no
Five Times Sit to Stand Test | Measurement at 12 weeks
  Part of short physical performance battery, yes vs no
Five Times Sit to Stand Test | Measurement at 24 weeks
  Part of short physical performance battery, yes vs no
Balance test | Measurement at discharge, baseline
  Part of short physical performance battery, yes vs no
Balance test | Measurement at 12 weeks
  Part of short physical performance battery, yes vs no
Balance test | Measurement at 24 weeks
  Part of short physical performance battery, yes vs no
Energy intake | Measurement at discharge, baseline
  Energy in kilocalories per 24 hours
Energy intake | Measurement at 12 weeks
  Energy in kilocalories per 24 hours
Energy intake | Measurement at 24 weeks
  Energy in kilocalories per 24 hours
Protein intake | Measurement at 12 weeks
  Protein intake in g/day
Protein intake | Measurement at discharge, baseline
  Protein intake in g/day
Protein intake | Measurement at 24 weeks
  Protein intake in g/day
Fluid intake | Measurement at discharge, baseline
  Fluid intake evaluated
Fluid intake | Measurement at 12 weeks
  Fluid intake evaluated
Fluid intake | Measurement at 24 weeks
  Fluid intake evaluated
Upper arm circumference | Measurement at discharge, baseline
  Measured in centimeters
Upper arm circumference | Measurement at 24 weeks
  Measured in centimeters
Waist circumference | Measurement at discharge, baseline
  Measured in centimeters
Waist circumference | Measurement at 24 weeks
  Measured in centimeters
calf circumference | Measurement at discharge, baseline
  Measured in centimeters
calf circumference | Measurement at 24 weeks
  Measured in centimeters
lean body mass | Measurement at discharge, baseline
  Measured with BIA (kg)
lean body mass | Measurement at 24 weeks
  Measured with BIA (kg)
Grip strength | Measurement at discharge, baseline
  Measured in kg
Grip strength | Measurement at 12 weeks
  Measured in kg
Grip strength | Measurement at 24 weeks
  Measured in lbs
Health Related Quality of Life (HRQL) | Measurement at discharge, baseline
  EQ-5D including SRH
Health Related Quality of Life (HRQL) | Measurement at 12 weeks
  EQ-5D including SRH
Health Related Quality of Life (HRQL) | Measurement at 24 weeks
  EQ-5D including SRH
Depression | Measurement at discharge, baseline
  Center for Epidemiologic Studies Depression scale
Depression | Measurement at 24 weeks
  Center for Epidemiologic Studies Depression scale
Cognitive function | Measurement at discharge, baseline
  MMSE
Cognitive function | Measurement at 24 weeks
  MMSE
Nutrition status | Measurement at discharge, baseline.
  Icelandic Nutrition Screening Tool (score)
Nutrition status | Measurement at 24 weeks
  Icelandic Nutrition Screening Tool (score)

SECONDARY OUTCOMES:
Re-hospitalization | at 12 months from recruitment to trial
  Number of participants who were re-hospitalized
Mortality | at 12 months from recruitment to trial
  Number of participants who deceased

CONTACTS AND LOCATIONS:
Overall Officials: Alfons Ramel, Ph.D., Principal Investigator — University of Iceland; Olof G Geirsdottir, Ph.D., Principal Investigator — University of Iceland; Berglind S Blondal, MSc, Principal Investigator — University of Iceland
Locations (1):
- Geriatric Unit of Landspitali - University Hospital of Iceland, Reykjavik, Non-US, Iceland

REFERENCES:
- [Derived] Eymundsdottir H, Blondal BS, Geirsdottir OG, Ramel A. Poor Activities of Daily Living Predict Future Weight Loss in Older Adults After Hospital Discharge-Secondary Analysis of a Randomized Trial. J Aging Phys Act. 2024 Aug 16;33(1):42-50. doi: 10.1123/japa.2023-0104. Print 2025 Feb 1. PMID 39151910
- [Derived] Blondal BS, Geirsdottir OG, Beck AM, Halldorsson TI, Jonsson PV, Sveinsdottir K, Ramel A. HOMEFOOD randomized trial-beneficial effects of 6-month nutrition therapy on body weight and physical function in older adults at risk for malnutrition after hospital discharge. Eur J Clin Nutr. 2023 Jan;77(1):45-54. doi: 10.1038/s41430-022-01195-2. Epub 2022 Aug 26. PMID 36028775